CLINICAL TRIAL: NCT01679418
Title: Randomized Controlled Trial on the Impact of Postoperative Drainage on Nausea and Vomiting After Thyroid- and Parathyroid Surgery
Brief Title: Impact of Drains on Postoperative Nausea and Vomiting After Thyroid Surgery
Acronym: PONTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Liestal (Other)
Responsible Party: Principal Investigator, Christoph A. Maurer, MD, Principal investigator, Kantonsspital Liestal
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PONV_thyroidsurgery
Record Dates: First submitted 2012-06-12; First posted 2012-09-06 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; thyroid; surgery; nausea and vomiting; postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Thyroid Diseases; Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drain placement (Group A) (Active Comparator): Patients in group A received a wound drain after surgery.
  Interventions: Device: Placement of a wound drain post surgery (Redon; Medicoplast)
- No-drain placement (group B) (Sham Comparator): Patients assigned to group B, did not receive a wound drain after surgery.
  Interventions: Other: No-drain after surgery

INTERVENTIONS:
Device: Placement of a wound drain post surgery (Redon; Medicoplast) — The wound drain, type Redon Drainage 3.0 mm in diameter
  Other Names: Redon Drainage (Ref. 750), 3.0 mm in diameter; Medicoplast, 66557 Illingen, Germany
  Arms: Drain placement (Group A)
Other: No-drain after surgery — After surgery, no drain was put
  Arms: No-drain placement (group B)

SUMMARY:
Wound Drains after Thyroid- and Parathyroid Surgery Impact on Postoperative Nausea and Vomiting (PONV)

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is common after thyroid surgery. Many patients describe PONV as more irritant in the postoperative course than the endured pain. Postoperative drains are put after thyroid surgery to early recognize bleeding and to collect wound secretion to avoid pressure on the trachea. Whether wound drains do impact on PONV is not known. Therefore, we tested the impact of wound drains on PONV after thyroid- and parathyroid surgery in a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years of age
* informed consent
* planed thyroid- or parathyroid resection
* euthyreostatic preoperative condition

Exclusion Criteria:

* younger than 18 years of age
* pregnancy
* no informed consent
* retrosternal struma
* known postoperative nausea and vomiting prior to surgery
* severe and life threatening systemic health issues

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assessment of post-operative nausea using visual analogue scale (VAS) | 24 hours post surgery
  The development of postoperative nausea was determined using a standard visual analogue scale (VAS) with range of 0 to 10. 0 indicated no nausea, 10 indicated very severe nausea. The patients indicated their felt degree of nausea a number between 0 to 10.
Assessment of postoperative vomiting using visual analogue scale (VAS) | 24 hours post surgery
  The development of postoperative vomiting was determined using a standard Visual analogue scale (VAS) with range of 0 to 10. 0 indicated no nausea, 10 indicated very severe nausea. The patients indicated their felt degree of vomiting indicating a number between 0 to 10. The number of vomiting was counted within the first 48h post surgery
Assessment of post-operative nausea using visual analogue scale (VAS) | 48 hours post surgery
  The development of postoperative nausea was determined using a standard visual analogue scale (VAS) with range of 0 to 10. 0 indicated no nausea, 10 indicated very severe nausea. The patients indicated their felt degree of nausea a number between 0 to 10.
Assessment of postoperative vomiting using visual analogue scale (VAS) | 48 hours post surgery
  The development of postoperative vomiting was determined using a standard Visual analogue scale (VAS) with range of 0 to 10. 0 indicated no nausea, 10 indicated very severe nausea. The patients indicated their felt degree of vomiting indicating a number between 0 to 10. The number of vomiting was counted within the first 48h post surgery

SECONDARY OUTCOMES:
Antiemetic therapy post surgery in patients with and without postoperative drainage | after 48 hours
  In the postoperative course, we counted the amount of anti-emetic interventions for patients post surgery over the first 48 hours. The givage of anti-emetic drugs was based on a prior determined protocol, that was strictly followed.
  The protocol was as follows for antiemetic drugs:
  First line Drug: Tropisetron 2 mg i.v. when patient is vomiting, max. twice a day. Second line therapy: Haloperidol 0.5 mg i.v. with a maximum of 3 mg every 24 hours, when first line therapy is not sufficient. The change to second line therapy is controlled by the study physician.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Maurer, MD, Study Director — Professor of Surgery, Head of the Department, Kantonsspital Liestal
Locations (1):
- Kantonsspital Liestal, Liestal, Basel-Landschaft, Switzerland

REFERENCES:
- [Background] Schwarz W, Willy C, Ndjee C. [Gravity or suction drainage in thyroid surgery? Control of efficacy with ultrasound determination of residual hematoma]. Langenbecks Arch Chir. 1996;381(6):337-42. doi: 10.1007/BF00191314. German. PMID 9082107
- [Derived] Kunzli BM, Walensi M, Wilimsky J, Bucher C, Buhrer T, Kull C, Zuse A, Maurer CA. Impact of drains on nausea and vomiting after thyroid and parathyroid surgery: a randomized controlled trial. Langenbecks Arch Surg. 2019 Sep;404(6):693-701. doi: 10.1007/s00423-019-01799-6. Epub 2019 Jun 26. PMID 31243574